CLINICAL TRIAL: NCT00466076
Title: Subcutaneous Copaxone as Treatment for Dry Age Related Macular Degeneration
Brief Title: Copaxone in Age Related Macular Degeneration
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kmc060033
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Macular Degeneration
Keywords: Drusen; AMD; Dry form of Age related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Copaxone (Glatiramer acetate)

SUMMARY:
The purpose of the project is to investigate in eyes with dry AMD, the efficacy and safety as preventive therapy of the immunomodulatory substance named copaxone which had been proven as safe and effective agent for a neurodegenerative disease, in arresting the progression as well as the conversion of dry AMD to wet AMD. The hypothesis that the immunomodulatory agent copaxone proven for a neurodegenerative disease may work in the eye is revolutionary and may open a new avenue of preventive treatment for the disease which is the major cause of legal blindness in the industrial world

DETAILED DESCRIPTION:
The formation of insoluble extracellular deposits consisting of misfolded, aggregated protein is the hallmark of many neurodegenerative diseases. Age-related macular degeneration (AMD) is a degenerative disease in the eye associated with extracellur deposits named drusen. Recent evidence suggests that drusen formation and AMD share some similarities with another neurodegenerative disease named Alzheimer's disease (AD) which is associated with amyloid deposits. AMD and AD are strongly correlated with advancing age and the formation of amyloid deposits. In addition, inflammatory mediators and in particular activated microglia are present in amyloid deposits as well as in drusen, suggesting a possible common role for the inflammatory pathway in AMD and amyloid diseases. Moreover, Ambati et al described a new model of AMD in transgenic mice when an absence of normally functioning macrophages led to the development of clinical AMD.

Michal Schwartz and her group have recently shown that aggregated b-amyloid (Ab) induces microglia to become cytotoxic and block neurogenesis from adult rodent neural progenitor cells (NPCs). IL-4, reversed the impediment, attenuated TNF-a production and overcame blockage of insulin like growth factor (IGF)-I production caused by Ab. The significance of microglia for in-vivo neural cell renewal was demonstrated by enhanced neurogenesis in the rat dentate gyrus after injection of IL-4-activated microglia intracerebroventricularly and by the presence of IGF-I-expressing microglia in the dentate gyrus of rats kept in an enriched environment or in the animal model of multiple sclerosis (MS). Using double-transgenic mice expressing mutant human genes encoding presenilin 1 and chimeric mouse/human amyloid precursor protein (mice Alzheimer's disease model), the group of Michal Schwartz showed that modulation of microglia into dendritic-like cells, achieved by a T cell-based vaccination with Copolymer-1 (Copaxone), resulted in reduction of cognitive decline, elimination of plaque formation, and induction of neuronal survival and neurogenesis. These results introduce a new microglia phenotype as necessary players in fighting off neurodegenerative conditions such as AD and AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Dry AMD in both eyes
2. Age 50 or above.
3. Signed informed consent.

Exclusion Criteria:

1. Known sensitivity to mannitol or Copaxone.
2. Skin disease or active infection of skin.
3. Active fever or active treatment for infection.
4. History of other active disaese.
5. Premenapausal females not using relibale birth control.
6. Sensitivity for flourescein or iodine.
7. Inability to comply with study procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-08; Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Total drusen area reduction

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Pollack, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Department of Ophthalmology, Kaplan Medical Center, Rehovot, Israel